CLINICAL TRIAL: NCT02717663
Title: WalkIT: Neighborhood Walkability and Moderation of Adaptive Walking Interventions
Brief Title: WalkIT Arizona: Walking Interventions Through Texting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marc Adams, PhD, MPH, Assistant Professor, Exercise and Wellness Program, School of Nutrition and Health Promotion, College of Health Solutions., Arizona State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01CA198915 (NIH); R01CA198915 (NIH)
Record Dates: First submitted 2016-03-10; First posted 2016-03-24 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Physical Activity; Behavior; Goals
Keywords: Reinforcement; Walking; Exercise; Built Environment; Adaptive; Financial incentive; Walkability
MeSH Terms: conditions — Motor Activity; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Static goals with delayed incentives (Experimental): Participants will receive static physical activity goals with delayed, non-contingent incentives
  Interventions: Behavioral: Static Goals; Behavioral: Delayed (non-contingent) Incentives
- Adaptive goals with delayed incentives (Experimental): Participants will receive adaptive physical activity goals with delayed, non-contingent incentives
  Interventions: Behavioral: Adaptive Goals; Behavioral: Delayed (non-contingent) Incentives
- Static goals with immediate rewards (Experimental): Participants will receive static physical activity goals with immediate rewards
  Interventions: Behavioral: Static Goals; Behavioral: Immediate Micro-Incentives
- Adaptive goals with immediate rewards (Experimental): Participants will receive adaptive physical activity goals with immediate rewards
  Interventions: Behavioral: Adaptive Goals; Behavioral: Immediate Micro-Incentives

INTERVENTIONS:
Behavioral: Adaptive Goals — Prescribed goals change daily based on participant's performance
  Arms: Adaptive goals with delayed incentives; Adaptive goals with immediate rewards
Behavioral: Static Goals — Prescribed goals remain the same throughout study
  Arms: Static goals with delayed incentives; Static goals with immediate rewards
Behavioral: Delayed (non-contingent) Incentives — Incentives are provided on bi-monthly basis for participation
  Arms: Adaptive goals with delayed incentives; Static goals with delayed incentives
Behavioral: Immediate Micro-Incentives — Incentives are provided immediately for each goal attained
  Arms: Adaptive goals with immediate rewards; Static goals with immediate rewards

SUMMARY:
The purpose of this study is to develop adaptive (AI) and micro-incentive (MI) interventions and test them against static (SI) and delayed-incentive (DI) interventions in a 4-arm randomized factorial trial to increase MVPA adoption and maintenance among inactive adults. Using neighborhood walkability and socioeconomic status, participants will be recruited from four neighborhood types: "high walkable/high SES," "high walkable/low SES," "low walkable/high SES," and "low walkable/low SES." We will evaluate synergistic or antagonistic effects of interventions and neighborhood factors on MVPA adoption by 12 months and maintenance by 24 months.

ELIGIBILITY:
Inclusion Criteria:

* women and men of all races/ethnicities living in Maricopa County, Arizona

Exclusion Criteria:

* Live in one of the eligible neighborhood quadrants in Maricopa County, Arizona
* Adult men and women between 18 and 60 years old
* Inactive as screened by the International Physical Activity Questionnaire (IPAQ) short form and confirmed by baseline accelerometer measures
* No history of heart failure or type 2 diabetes
* No contraindications to exercise testing or requirement for medically supervised exercise (assessed by Physical Activity Readiness Questionnaire+ (PAR-Q+).
* Not currently pregnant and not planning to becoming pregnant in the next 2 years
* Not currently participating in physical activity, diet, or weight loss programs
* Daily access to a mobile phone with text messaging capabilities or an iOS or Android smartphone
* Willing to wear a small accelerometer on the wrist daily for 1 year
* Willing to send and receive 2-3 text messages per day for 1 year
* Not planning to be outside of Maricopa County for > 30 days consecutively in the next 2 years
* Not planning to move from their current home in the next 2 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 512 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Change in mean ActiGraph accelerometer-derived moderate-to-vigorous physical activity min/day (MVPA min/day) between study arms. | 12 months
Change in mean ActiGraph accelerometer-derived moderate-to-vigorous physical activity min/day (MVPA min/day) across high walkable (vs. low walkable) neighborhoods by 12 months. | 12 months
Change in mean ActiGraph accelerometer-derived moderate-to-vigorous physical activity min/day (MVPA min/day) across high walkable (vs. low walkable) neighborhoods by 24 months | 24 months

SECONDARY OUTCOMES:
Change in mean fitness (VO2max measured by treadmill test) between study arms. | 12 months
Change in self-reported physical activity measured by the International Physical Activity Questionnaire (IPAQ). | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McEntee ML, Hurley JC, Phillips CB, Hooker SP, Todd M, Frank LD, Adams MA. The moderating impact of neighborhood walkability on mHealth interventions to increase moderate to vigorous physical activity for insufficiently active adults in a randomized trial. Int J Behav Nutr Phys Act. 2023 Aug 15;20(1):97. doi: 10.1186/s12966-023-01494-2. PMID 37582736
- [Derived] Adams MA, Todd M, Angadi SS, Hurley JC, Stecher C, Berardi V, Phillips CB, McEntee ML, Hovell MF, Hooker SP. Adaptive Goals and Reinforcement Timing to Increase Physical Activity in Adults: A Factorial Randomized Trial. Am J Prev Med. 2022 Feb;62(2):e57-e68. doi: 10.1016/j.amepre.2021.09.014. Epub 2021 Dec 8. PMID 35000693
- [Derived] McEntee ML, Cantley A, Foreman E, Berardi V, Phillips CB, Hurley JC, Hovell MF, Hooker S, Adams MA. Effects of Goal Type and Reinforcement Type on Self-Reported Domain-Specific Walking Among Inactive Adults: 2x2 Factorial Randomized Controlled Trial. JMIR Form Res. 2020 Dec 4;4(12):e19863. doi: 10.2196/19863. PMID 33275107